CLINICAL TRIAL: NCT03166020
Title: Evaluation of a Video-ludic Re-education of the Paretic Upper Limb in Chronic Hemipartic Patients Post Cerebral Vascular Accident
Acronym: ERGOTACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: Fondation Garches (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-A01903-48
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2018-05

CONDITIONS: Stroke; Motor Activity
Keywords: Serious Game; Stroke; Rehabilitation; Connected objects
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation with Interactive Table (Experimental): Included patients will be invited to participate in 10 sessions, focused on the movement and manipulation of instrumented objects on interactive table with serious game, during 30 minutes per day, 5 days a week, for 14 days. An occupational therapist will be required only for patient installation in front of the table.
  Interventions: Other: Rehabilitation
- Self Rehabilitation (Active Comparator): Included patients will be instructed to perform 10 self-rehabilitation sessions with 9 exercises (3 stretching, 3 reinforcement, 3 spot-oriented work) during 30 minutes per day, 5 days a week, for 14 days.
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — An occupational therapist will be required only for patient installation in front of the table.

SUMMARY:
The aim of this randomized controlled study with stroke patients is to demonstrate that a re-education with interactive table with instrumented objects delivering sensory feedback and serious game improve certain motor functions of the paretic upper limb than rehabilitation based on a standardized self-rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients
* Subject with gripping ability: capable of peeling off the connected object from the table, presented in its grip area.

Exclusion Criteria:

* Severe cognitive disorders preventing the completion of the task
* Bilateral brain lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
Speed of the gesture to reach each target | 10 minutes
  score

SECONDARY OUTCOMES:
Wolf Motor Functional Test | 15 minutes
  Clinical Evaluation
Box and block | 5 minutes
  Clinical Evaluation
Fugl Meyer | 10 minutes
  Clinical Evaluation
MOCA | 5 minutes
  Clinical Evaluation
Pain | 1 minute
  Visual analog scale
Spasticity | 5 minutes
  Visual analog scale
SF12 Quality of life | 10 minutes
  Clinical Evaluation
Canadian Occupational Performance Measure | 20 minutes
  Clinical Evaluation
Frenchay activities Index | 15 minutes
  Clinical Evaluation
Cinematic Evaluation | 10 minutes
  Evaluation of the cinematic of the paretic upper limb
Clamping force | 2 minutes
  composite score

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas ROCHE, MD phD, Principal Investigator — Raymond Poincare HOSPITAL
Locations (2):
- France (2):
  - Hopital Raymond Poincare, Garches
  - Nicolas ROCHE, Md PhD, Garches

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pouplin S, Bonnyaud C, Bouchigny S, Megard C, Bertholier L, Goulamhoussen R, Foulon P, Bensmail D, Barbot F, Roche N. Feasibility of a serious game system including a tangible object for post stroke upper limb rehabilitation: a pilot randomized clinical study. Front Neurol. 2023 Jun 9;14:1176071. doi: 10.3389/fneur.2023.1176071. eCollection 2023. PMID 37360348